CLINICAL TRIAL: NCT06188195
Title: Establishment and Evaluation of Prenatal Prevention and Treatment Strategy for Neonatal Acute Respiratory Distress Syndrome
Brief Title: Establishment and Evaluation of Prenatal Prevention and Treatment Strategy for NARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: University-Town Hospital of Chongqing Medical University (Other); Children's Hospital of Chongqing Medical University (Other); Chongqing Medical Center for Women and Children (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LWang
Record Dates: First submitted 2023-11-27; First posted 2024-01-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-12

CONDITIONS: Acute Respiratory Distress Syndrome; Respiratory Distress Syndrome, Acute
Keywords: Neonatal Acute Respiratory Distress Syndrome; Prediction nomogram; antenatal corticosteroids
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the experimental group (Experimental): For pregnant women with a probability greater than 80% in the prediction model of NARDS, those who agreed to ACS intervention were included in the experimental group
  Interventions: Drug: Dexamethasone
- the control group (No Intervention): For pregnant women with a probability greater than 80% in the prediction model of NARDS, those who did not agree with ACS intervention were included in the control group

INTERVENTIONS:
Drug: Dexamethasone — ACS intervention were used in the experimental group
  Other Names: antenatal corticosteroids
  Arms: the experimental group

SUMMARY:
1. A predictive model for NARDS was established based on perinatal risk factors. Multivariate Logistic regression analysis was used to screen the independent prenatal risk factors for NARDS. A Logistic regression model was constructed using the above independent risk factors and quantified in a nomogram to construct a visualization model for prenatal prediction of NARDS.
2. The role of ACS in the prevention and treatment of ARDS in near-term/full-term infants.

For neonates with a probability greater than 80% in the prediction model of ARDS, at least one ACS was given before the termination of pregnancy. The GC level of cord blood (taken at birth) and the mRNA levels of α-ENaC, Na-K-atpase and SGK1 in nasal epithelium were measured within 2 hours and 1 day after birth in the ACS intervention group and the control group. The occurrence and severity of pulmonary edema, the occurrence and severity of ARDS, and the mortality rate of NARDS were evaluated by lung ultrasound. The indexes of the two groups were compared horizontally and longitudinally.

DETAILED DESCRIPTION:
Based on the proposed scientific hypothesis, the project team intends to achieve the following research objectives through scientific experiments:

To explore the role of ACS in promoting fetal lung maturation from the perspective of lung fluid clearance through the traditional concept that ACS promotes fetal lung maturation mainly by inducing PS, so as to further expand the object and scope of ACS application.

The prenatal prediction model of ARDS was established by using perinatal risk factors, and the predictive value was visualized.

To explore the clinical value and mechanism of ACS in pregnant women at high risk of NARDS, and to open up new ideas for the prevention and treatment of NARDS from the perspective of promoting lung fluid clearance; The early prevention and treatment strategy of NARDS was established by combining the "prenatal prediction model +ACS", and its effect was evaluated.

ELIGIBILITY:
A predictive model for neonatal acute respiratory distress syndrome was established based on perinatal risk factors.

Inclusion Criteria:

1. The pregnant women with a probability greater than 80% in the prediction model of neonatal acute respiratory distress syndrome and agreed to ACS intervention.
2. Obtaining patient consent.

Exclusion Criteria:

1. the pregnant women with a probability of less than 80% in the neonatal acute respiratory distress syndrome prediction model.
2. The patient refuses.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of neonatal acute respiratory distress syndrome | 1 year
  The incidence and severity of neonatal acute respiratory distress syndrome will be compared between the two groups
The incidence and severity of pulmonary edema | 1 year
  The incidence and severity of pulmonary edema will be compared between the two groups
The mortality of NARDS | 1 year
  The mortality rate of NARDS will be compared between the two groups
The mRNA levels of α-ENaC, Na-K-atpase, and SGK1 in nasal epithelium | Day 0 after birth
  The mRNA levels of α-ENaC, Na-K-atpase, and SGK1 in nasal epithelium will be compared between the two groups
The glucocorticoid level in cord blood | Day 0 after birth
  The glucocorticoid levels of cord blood will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Li Wang, MD,PhD, Study Chair — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Luca D, van Kaam AH, Tingay DG, Courtney SE, Danhaive O, Carnielli VP, Zimmermann LJ, Kneyber MCJ, Tissieres P, Brierley J, Conti G, Pillow JJ, Rimensberger PC. The Montreux definition of neonatal ARDS: biological and clinical background behind the description of a new entity. Lancet Respir Med. 2017 Aug;5(8):657-666. doi: 10.1016/S2213-2600(17)30214-X. Epub 2017 Jul 4. PMID 28687343
- [Background] Wang L, Chen L, Li R, Zhao J, Wu X, Li X, Shi Y. Efficacy of surfactant at different gestational ages for infants with respiratory distress syndrome. Int J Clin Exp Med. 2015 Aug 15;8(8):13783-9. eCollection 2015. PMID 26550326
- [Background] Cantarutti A, Franchi M, Monzio Compagnoni M, Merlino L, Corrao G. Mother's education and the risk of several neonatal outcomes: an evidence from an Italian population-based study. BMC Pregnancy Childbirth. 2017 Jul 12;17(1):221. doi: 10.1186/s12884-017-1418-1. PMID 28701151
- [Background] Venkatesh KK, Jackson W, Hughes BL, Laughon MM, Thorp JM, Stamilio DM. Correction: Association of chorioamnionitis and its duration with neonatal morbidity and mortality. J Perinatol. 2019 May;39(5):761. doi: 10.1038/s41372-019-0341-x. PMID 30842550
- [Background] Liu H, Li J, Guo J, Shi Y, Wang L. A prediction nomogram for neonatal acute respiratory distress syndrome in late-preterm infants and full-term infants: A retrospective study. EClinicalMedicine. 2022 Jun 25;50:101523. doi: 10.1016/j.eclinm.2022.101523. eCollection 2022 Aug. PMID 35784441
- [Background] Polnaszek B, Lopez JD, Clark R, Raghuraman N, Macones GA, Cahill AG. Marked variability in intrapartum electronic fetal heart rate patterns: association with neonatal morbidity and abnormal arterial cord gas. J Perinatol. 2020 Jan;40(1):56-62. doi: 10.1038/s41372-019-0520-9. Epub 2019 Oct 2. PMID 31578422
- [Background] Suvari L, Helve OM, Kari MA, Turpeinen LU, Palojarvi PA, Leskinen MJ, Andersson S, Janer AC. Glucocorticoids, sodium transport mediators, and respiratory distress syndrome in preterm infants. Pediatr Res. 2021 Apr;89(5):1253-1260. doi: 10.1038/s41390-020-1061-9. Epub 2020 Jul 14. PMID 32663837
- [Background] Saccone G, Berghella V. Antenatal corticosteroids for maturity of term or near term fetuses: systematic review and meta-analysis of randomized controlled trials. BMJ. 2016 Oct 12;355:i5044. doi: 10.1136/bmj.i5044. PMID 27733360
- [Background] Smith GC. Antenatal Betamethasone for Women at Risk for Late Preterm Delivery. N Engl J Med. 2016 Aug 4;375(5):486. doi: 10.1056/NEJMc1605902. No abstract available. PMID 27518672
- [Background] Sheibani L, Fong A, Henry DE, Norton ME, Truong YN, Anyikam A, Laurent LC, Rao R, Wing DA; University of California Fetal Consortium (UCfC). Maternal and neonatal outcomes after antenatal corticosteroid administration for PPROM at 32 to 33 6/7 weeks gestational age. J Matern Fetal Neonatal Med. 2017 Jul;30(14):1676-1680. doi: 10.1080/14767058.2016.1222366. Epub 2016 Aug 31. PMID 27578238
- [Background] Amiya RM, Mlunde LB, Ota E, Swa T, Oladapo OT, Mori R. Antenatal Corticosteroids for Reducing Adverse Maternal and Child Outcomes in Special Populations of Women at Risk of Imminent Preterm Birth: A Systematic Review and Meta-Analysis. PLoS One. 2016 Feb 3;11(2):e0147604. doi: 10.1371/journal.pone.0147604. eCollection 2016. PMID 26841022
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GH, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2016 Update. Neonatology. 2017;111(2):107-125. doi: 10.1159/000448985. Epub 2016 Sep 21. PMID 27649091
- [Background] Miyazaki K, Furuhashi M, Ishikawa K, Tamakoshi K, Hayashi K, Kai A, Ishikawa H, Murabayashi N, Ikeda T, Kono Y, Kusuda S, Fujimura M. Long-term outcomes of antenatal corticosteroids treatment in very preterm infants after chorioamnionitis. Arch Gynecol Obstet. 2015 Dec;292(6):1239-46. doi: 10.1007/s00404-015-3762-6. Epub 2015 May 20. PMID 25990481